CLINICAL TRIAL: NCT05584839
Title: A Comprehensive Statistical Analysis for the Diagnosis of Carpal Tunnel Syndrome
Brief Title: Statistically Analysis of Carpal Tunnel Syndrome Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: İSMAİL CEYLAN (Other)
Responsible Party: Sponsor-Investigator, İSMAİL CEYLAN, Head of hand therapy clinic. PhD., Ahi Evran University Education and Research Hospital
Organization: Ahi Evran University Education and Research Hospital (Other)
Other Study IDs: 12068451745
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Carpal Tunnel Syndrome; Diagnosis
Keywords: carpal tunnell syndrome; anthpometric
MeSH Terms: conditions — Carpal Tunnel Syndrome; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- carpal tunnel syndrome: * Admitted to outpatient clinics with symptoms of CTS
  * Findings of CTS in physical examination
  * CTS diagnosis was confirmed by nerve conduction study
  * KTS grade mild or moderate
  * He has not received physical therapy for this reason in the previous 1 year
  * No steroid injection and no treatment for neuropathic pain (pregabalin, gabapentin, etc.)
  Interventions: Other: Statistically Analysis

INTERVENTIONS:
Other: Statistically Analysis — The study was planned as a quantitative research. Socio-demographic information form, anthropometric measurements of hand grip strength, palm length, hand width length, wrist circumference length, Visual Analog Scale scale, EMG findings will be evaluated by hand dynamometer.

SUMMARY:
Trap neuropathies; They are compression neuropathies that occur as a result of peripheral nerves being compressed for various reasons along their anatomical paths. Although each nerve has areas suitable for anatomical entrapment, compression can occur at any point along the nerve. Carpal tunnel syndrome (CTS) is the most common entrapment neuropathy caused by compression of the median nerve at the wrist level. Its prevalence in the general population is 2.5-11%.

Although the majority of cases are idiopathic, it may also occur secondary to pathologies such as pregnancy, diabetes mellitus, thyroid dysfunction, arthritis, wrist fractures and acromegaly or occupation. The diagnosis of CTS is made clinically, but the best method for definitive diagnosis is electrophysiological examination.

Some anthropometric measurements that may be associated with CTS were made and their effect on the risk of CTS was investigated. In a study conducted by Sabry et al. in 2009, it was reported that there may be a relationship between BMI, wrist ratio (ratio of wrist depth to width) and wrist-palm ratio (ratio of wrist depth to palm length) and CTS risk. In a study by Lim et al. in 2008, it was reported that the critical value for wrist ratio was 0.70 and above. However, there were no studies reporting how many percent predictors of anthropometric measurements according to the severity of CTS.

DETAILED DESCRIPTION:
The study was planned as a quantitative research. Socio-demographic information form, anthropometric measurements of hand grip strength, palm length, hand width length, wrist circumference length, Visual Analog Scale scale, EMG findings will be evaluated by hand dynamometer.

Trybus et al. Considering the study they conducted in patients with CTS in which they examined hand anthropometric measurements in CTS, it was planned to include 100 patients in the study with a power range of 80% and an effect width of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to outpatient clinics with symptoms of CTS
* Findings of CTS in physical examination
* CTS diagnosis was confirmed by nerve conduction study
* KTS grade mild or moderate
* He has not received physical therapy for this reason in the previous 1 year
* No steroid injection and no treatment for neuropathic pain (pregabalin, gabapentin, etc.)

Exclusion Criteria:

* - Those under the age of 18 Those with a history of previous surgery or fracture of the affected hand and wrist Those with diabetes mellitus, chronic kidney failure, gout, rheumatoid arthritis, thyroid diseases
* Pregnant Those with polyneuropathy, radiculopathy, plexopathy, thoracic outlet syndrome

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Persons aged 18-65 years who apply to outpatient clinics with symptoms of CTS
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Hand Grip Strength | 0-1 days
  The grip strength of the dominant hand is measured using a standard adjustable digital grip dynamometer (Baseline Digital Smedley Hand Dynamometer). Handgrip strength is measured as follows: (a) Each subject is tested while sitting comfortably in a chair without armrests, with their back against the chair; (b) Each subject is instructed to sit with hips and knees flexed 90°, shoulders adducted and neutrally rotated, elbows flexed 90°, forearm rotation 0°, wrists dorsiflexed 0° to 30°, and ulnar deviation 0° to 15°; and asked to squeeze the dynamometer.

SECONDARY OUTCOMES:
Hand length | 0-1 days
  Hand length is moderate when forearm and hand are brought to supination on a table.
  is the distance from the tip of the finger to the midline of the distal wrist crease.

CONTACTS AND LOCATIONS:
Locations (1):
- İsmail Ceylan, Kırşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Calixtre LB, Oliveira AB, de Sena Rosa LR, Armijo-Olivo S, Visscher CM, Alburquerque-Sendin F. Effectiveness of mobilisation of the upper cervical region and craniocervical flexor training on orofacial pain, mandibular function and headache in women with TMD. A randomised, controlled trial. J Oral Rehabil. 2019 Feb;46(2):109-119. doi: 10.1111/joor.12733. Epub 2018 Oct 26. PMID 30307636